CLINICAL TRIAL: NCT02369107
Title: A Multi-center,Randomized Controlled Clinical Trial: the Effect of Acupuncture in Prevention and Treatment of Chemotherapy-induced Nausea and Vomiting on Patients With Malignancy
Brief Title: The Effect of Acupuncture in Chemotherapy-induced Nausea and Vomiting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Friendship Hospital (Other); Beijing Municipal Administration of Hospitals (Other Government)
Responsible Party: Principal Investigator, Wang Xiaomin, Doctor, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XM201410
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
Keywords: acupuncture; chemotherapy-induced nausea and vomiting
MeSH Terms: conditions — Vomiting | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum acupuncture and medicine (Experimental): Participants will receive acupuncture therapy 1 hour prior to chemotherapy administration ，6 hours after chemotherapy administration，and once acupuncture therapy on the following day2,3,4,5. The stimulation points are RN12,LR13(bilaterally), RN6, ST25(bilaterally), PC6(bilaterally), ST36(bilaterally). The acupuncture needle in ST36 and auxiliary point will be connected to form a circuit containing a SDZ-V stimulator for 30 min with a frequency of 2/100 Hz.They will receive 8mg Ondansetron Intravenously twice a day during the chemotherapy administration period (5 days in total).
  Interventions: Other: Verum acupuncture and medicine
- Sham acupuncture and medicine (Sham Comparator): Participants will receive minimal acupuncture therapy at the same time as the intervention group .The stimulation points are not belong to traditional Chinese medicine.They will receive 8mg Ondansetron Intravenously twice a day during the chemotherapy administration period (5 days in total).
  Interventions: Other: Sham acupuncture and medicine

INTERVENTIONS:
Other: Verum acupuncture and medicine — Participants will receive acupuncture therapy 1 hour prior to chemotherapy administration ，6 hours after chemotherapy administration，and once acupuncture therapy on the following day2,3,4,5. The stimulation points are RN12,LR13(bilaterally), RN6, ST25(bilaterally), PC6(bilaterally), ST36(bilaterally). The acupuncture needle in ST36 and auxiliary point will be connected to form a circuit containing a SDZ-V stimulator for 30 min with a frequency of 2/100 Hz. They will receive 8mg Ondansetron Intravenously twice a day during the chemotherapy administration period (5 days in total).
  Arms: Verum acupuncture and medicine
Other: Sham acupuncture and medicine — Participants will receive minimal acupuncture therapy at the same time as the intervention group .The stimulation points are not belong to traditional Chinese medicine.They will receive 8mg Ondansetron Intravenously twice a day during the chemotherapy administration period (5 days in total).
  Arms: Sham acupuncture and medicine

SUMMARY:
Nausea and vomiting are the most common symptoms experienced by cancer patients after chemotherapy. Some patients have to endure such unpleasant symptoms even after using of antiemetic or anti-vomiting medications.The purpose of this study is to assess the therapeutic effects and safety of acupuncture for chemotherapy-induced nausea and vomiting on patients with malignancy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with definite pathological diagnosis of lung cancer, breast cancer, and gynecological cancer.They haven't receive any chemotherapy or radiotherapy treatment for three months prior to join this study.
2. Aged 18-75.
3. Patients will receive chemotherapy treatment which included Cisplatin, anthracycline or taxane during the study period.
4. ECOG score is between 0 and 2.
5. The patients are diagnosed with insufficiency of spleen-qi and stomach-qi,reverse ascending of Stomach-Qi in traditional Chinese medicine theory.
6. The expected lifetime of the patient is longer than 6 months.
7. Patients willing to participate in the study and sign the consent form.

Exclusion Criteria:

1. Patients have serious disease in cardiovascular system ,liver system,kidney system, immune systems and hemopoietic system.
2. Pregnant and lactating women.
3. Patients have intractable vomiting caused by malignant brain metastases, intracranial hypertention, digestive tract obstruction, severe liver or Renal dysfunction, brain tumors, cerebrovascular disease, or other reasons.
4. Patients with Coagulopathy, thrombocytopenia, or suffering from bleeding disorders.
5. Patients have been definitely diagnosed with depression, anxiety disorders and psychosis
6. Patients with Sepsis or Bacteremia.
7. Patients have lymphedema in acupuncture stimulation area.
8. Patients who are afraid of acupuncture stimulation or allergic to stainless steel needles can't participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in severity of nausea and vomiting at 21 days | It will be assessed at baseline,day1, day 2, day 3, day 7(±1)，day 10(±1), day 14(±1), day 21(±1).Patients have a daily questionnaire about nausea and vomiting during chemotherapy to record their feelings
  The severity of nausea and vomiting will be assessed by the Common Terminology Criteria for Adverse Events (CTCAE)

SECONDARY OUTCOMES:
TCM symptoms scale | It will be assessed at baseline, day3, day7(±1), day14(±1), day21(±1).Patients will be accessed with questionaire by doctors.
  to evaluate TCM syndrome
ECOG score scale | It will be assessed at baseline, day3, day7(±1), day14(±1), day21(±1).Patients will be accessed with questionaire by doctors.
  to evaluate physical condition of patients
HADS | It will be assessed at baseline, day3, day7(±1), day14(±1), day21(±1).Patients will be accessed with questionaire by doctors.
  a questionnaire to access the anxiety levels of patients

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomin Wang, Doctor, Principal Investigator — Beijing Hospital of Traditional Chinese Medicine

REFERENCES:
- [Derived] Li QW, Yu MW, Yang GW, Wang XM, Wang H, Zhang CX, Xue N, Xu WR, Fu Q, Yang Z, Yang L. Effect of acupuncture in prevention and treatment of chemotherapy-induced nausea and vomiting in patients with advanced cancer: study protocol for a randomized controlled trial. Trials. 2017 Apr 20;18(1):185. doi: 10.1186/s13063-017-1927-2. PMID 28427442